CLINICAL TRIAL: NCT01604070
Title: Randomized Multi-Center Post Market Clinical Study to Evaluate the Safety and Performance of NextraTM for Use in Foot Surgery to Fuse the Proximal-interphalangeal- Joints
Brief Title: Study to Evaluate Safety, of NextraTM in Surgery to Fuse the Proximal-interphalangeal- Joints
Status: Completed | Type: Observational
Sponsor: eMedtrain Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Nextremity_2011
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Foot Diseases
Keywords: Hammertoe deformity; podiatry
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Nextra fusion: group that has the nextra device
- k wire fixation: control group fixated with k wire

SUMMARY:
Hammertoe deformity is the most common deformity of the lesser toes. It primarily comprises flexion deformity of the proximal interphalangeal (PIP) joint of the toe, with hyperextension of the metatarsophalangeal (MTP).

Etiologies of hammertoe deformity include a foot in which the second ray is longer than the first, MTP synovitis and instability, inflammatory arthropathies, neuromuscular conditions, and ill-fitting shoe wear. When a foot's second ray is longer than the first and shoe wear does not fit correctly, flexion of the PIP joint occurs to accommodate the shoe. This length difference also causes MTP synovitis to develop from overuse of the second MTP joint. Attenuation of the collateral ligaments and plantar plate result, and the MTP joint hyperextends and may even progress to dorsal subluxation or dislocation (see image below). Rheumatoid arthritis causes hammertoe deformity by progressive MTP joint destruction, leading to MTP joint subluxation and dislocation.

With all 3 of these etiologies, the extensor digitorum longus (EDL) tendon gradually loses mechanical advantage at the PIP joint, as does the flexor digitorum longus (FDL) tendon at the MTP joint. The intrinsic muscles fire and sublux dorsally, as the MTP hyperextends. They now extend the MTP joint and flex the PIP joint, as opposed to their usual functions of flexing the MTP joint and extending the PIP joint.

DETAILED DESCRIPTION:
Device Description:

Nextra implant is an anatomical 2-piece designed implant with 10° angulation with a locking fusion mechanism. The self-centering, metaphysis screw design allows a stable and secure relationship of the proximal and middle phalanges. The compression with progressive tightening approximates the bone surfaces for a controlled fusion.

Pre-clinical Data:

The Nextra Implant has been used to create fusions between the proximal and middle phalanges of the 2nd, 3rd. or 4th. toe.

Clinical Experience:

The NextraTM Implant has been used in humans as an implant to reduce hammertoe and contracture deformities.

2. STUDY OBJECTIVES: The primary objective is to evaluate the post-market safety and performance of NextraTM in the reduction of post-operative pain symptoms in hammertoes and demonstrate the efficacy of the implant to securely stabilize bone surfaces to be fused as to be compared to K-wire fixation.

3. STUDY DESIGN: General Design: Preoperative and post-operative factors will be assessed in the evaluation of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the toe reported for greater than 3 months.
* Subjects are males or females,
* Diagnosed with a hammertoe, contracture of the IPJ, or other condition,
* Requiring digital proximal inter-phalangeal joint fusion of the 2nd, 3rd or 4th toe.
* Unilateral deformity of a single digit (2nd, 3rd or 4th)
* Subjects will sign an informed consent.
* Subjects are willing to return for follow-up visits and fill out Quality of Life questionnaires

Exclusion Criteria:

* Previous digital fusion surgery Previous PIPJ arthroplasty
* Bilateral surgery Hallux valgus creating a crossover toe with 2nd toe
* Inability to walk without an assistive device
* Infection Rheumatic joint disease
* Peripheral vascular disease with sensory loss to the toe
* Pregnant
* Osteoporosis
* Obvious loss of digital bone density Severe respiratory disease
* Open wounds
* Patients presently taking Gabapentin (Neurontin), Pregabalin (Lyrica), etc. drugs for neuropathic pain
* Diabetics
* Narcotic dependence
* Inability to consent to the research
* Concurrent involvement in another clinical trial
* Known allergy to the device components
* Known metabolic bone disease
* Renal disease (CRI, CRF)
* Skeletal muscle spasticity or paralysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a post market study and will consist of patients meeting the inclusion and exclusion criteria. The investigator recruits subjects if they meet the Inclusion/Exclusion requirements and are willing to sign an Informed Consent. Since the product is commercially available, randomization will occur at the time of surgery. Randomization will be according to a randomization table provided to the site investigators. The Surgeon will be unblended, and the subject will be blinded as to his/ her group (Treated-implant or Control-pin fixation).
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
fusion | 6 months
  proximal phalanx fusion

SECONDARY OUTCOMES:
patient perception of outcome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rick Jay, DPM, Principal Investigator — Pennsylvania Hospital; Adam Landsman, DPM, Principal Investigator — Cambridge Hospital; Michael Trepal, DPM, Principal Investigator — Foot Clinics of New York; Nelson G Keller, DPM, Principal Investigator — Mary Immaculate Hospital; Phillip Garrett, DPM, Principal Investigator — Inova Alexandria Hospital
Locations (4):
- United States (4):
  - Cambridge Hospital, Cambridge, Massachusetts
  - Cumberland Orthopedic, Vineland, New Jersey
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Mary Immaculate Hospital, Newport News, Virginia